CLINICAL TRIAL: NCT07175493
Title: A Phase 1/2 Clinical Study of CM336 Injection in Patients With Relapsed or Refractory Autoimmune Cytopenia
Brief Title: A Study of CM336 in Patients With Relapsed or Refractory Autoimmune Cytopenia
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Keymed Biosciences Co.Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CM336-125101
Record Dates: First submitted 2025-08-29; First posted 2025-09-16 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Autoimmune Cytopenia; Immune Thrombocytopenia (ITP); Autoimmune Hemolytic Anemia; Evans Syndrome
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Anemia, Hemolytic, Autoimmune; Evans Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CM336 injection (Experimental)
  Interventions: Biological: CM336 Injection

INTERVENTIONS:
Biological: CM336 Injection — subcutaneous CM336 administration, step-up dosing, Dose and frequency of CM336 according to the protocol

SUMMARY:
To evaluate the efficacy and safety of CM336 (BCMA/CD3 Bispecific Antibody) in the treatment of patients with relapsed or refractory autoimmune cytopenia

ELIGIBILITY:
Inclusion Criteria:

* Voluntary provision of written informed consent and ability to comply with protocol requirements.
* Age ≥18 years, male or female.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 2.
* Confirmed diagnosis of immune thrombocytopenia (ITP), warm autoimmune hemolytic anemia (wAIHA), cold agglutinin disease (CAD), mixed autoimmune hemolytic anemia (mAIHA) or Evans Syndrome.
* Relapsed or refractory autoimmune hemolytic anemia.

Exclusion Criteria:

* Secondary ITP or AIHA caused by any reason. Subjects with positive autoimmune antibodies but without a clear diagnosis of any other autoimmune diseases are allowed to be enrolled.
* Other types of AIHA or other types of cytopenia
* History of critical diseases that, in the opinion of the investigator, may pose a risk to the safety of subjects or whose exacerbation during the study could compromise the efficacy or safety analysis of the results.
* Received any treatment of anti-B Cell Maturation Antigen(BCMA) antibody.
* Evaluated unsuitable to participant in this study by investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2025-11-18 (Actual); Primary Completion 2027-11-18 (Estimated); Study Completion 2028-11-18 (Estimated)

PRIMARY OUTCOMES:
Incidence and Severity of Adverse Events (AEs) and Serious Adverse Events (SAEs) | 52 weeks
  Safety will be assessed by monitoring the incidence, nature, and severity of treatment-emergent adverse events (TEAEs), including serious adverse events (SAEs), adverse events of special interest (AESIs) such as cytokine release syndrome (CRS) and immune effector cell-associated neurotoxicity syndrome (ICANS), graded according to NCI CTCAE v5.0 and American Society for Transplantation and Cellular Therapy(ASTCT) criteria. Dose interruptions, modifications, or discontinuations due to toxicity will also be recorded.
Efficacy of CM336 | 8 weeks
  Overall hematological response rate within 8 weeks
Proportion of ITP subjects with a platelet count ≥ 50 × 10^9/L at least twice during the visit. | up to 52 weeks.
  Proportion of ITP subjects with a platelet count ≥ 50 × 10^9/L at least twice during the visit.
Proportion of AIHA subjects with at least one instance of hemoglobin ≥ 100 g/L, and an increase ≥ 20 g/L compared to the baseline level. | up to 52 weeks.
  Proportion of AIHA subjects with at least one instance of hemoglobin ≥ 100 g/L, and an increase ≥ 20 g/L compared to the baseline level.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Heping Hospital Affiliated to Changzhi Medical College, Changzhi, Shanxi
  - Blood Disease Hospital, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality